CLINICAL TRIAL: NCT03092323
Title: SU2C-SARC032: A Phase II Randomized Controlled Trial of Neoadjuvant Pembrolizumab With Radiotherapy and Adjuvant Pembrolizumab in Patients With High-Risk, Localized Soft Tissue Sarcoma of the Extremity
Brief Title: A Randomized Trial of Pembrolizumab & Radiotherapy Versus Radiotherapy in High-Risk Soft Tissue Sarcoma of the Extremity
Acronym: SU2C-SARC032
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sarcoma Alliance for Research through Collaboration (Other)
Collaborators: Stand Up To Cancer (Other); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SU2C-SARC032
Record Dates: First submitted 2017-03-15; First posted 2017-03-27 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-05

CONDITIONS: Soft Tissue Sarcoma of the Extremity
MeSH Terms: interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Neoadjuvant pembrolizumab with concurrent radiotherapy, followed by surgical resection and adjuvant pembrolizumab.
  Interventions: Drug: Pembrolizumab
- Standard of Care (No Intervention): Neoadjuvant radiotherapy followed by surgical resection.

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab will be administered at 200 mg intravenously every 3 weeks for patients on the treatment arm.
  Other Names: KEYTRUDA®
  Arms: Treatment

SUMMARY:
This is an open-label, multi-institutional phase II randomized study comparing neoadjuvant radiotherapy followed by surgical resection to neoadjuvant pembrolizumab with concurrent radiotherapy, followed by surgical resection and adjuvant pembrolizumab. The total duration of pembrolizumab will be one year in the experimental arm.

DETAILED DESCRIPTION:
This is a multicenter, randomized phase II trial with an initial safety run-in to test the safety and efficacy of neoadjuvant pembrolizumab with image-guided radiotherapy and adjuvant pembrolizumab compared to radiation therapy alone in patients with clinically localized extremity soft tissue sarcoma at high risk for developing metastatic disease (tumor size > 5 cm, intermediate- to high-grade; approximately 50% risk for distant disease at 2 years). Histologies will be limited to undifferentiated pleomorphic sarcoma and dedifferentiated/pleomorphic liposarcoma based on preliminary data from SARC028. Other terms for undifferentiated pleomorphic sarcoma may include, but are not limited to. pleomorphic undifferentiated sarcoma, unclassified spindle cell sarcoma, spindle cell sarcoma not otherwise specified, pleomorphic spindle cell sarcoma, pleomorphic fibroblastic sarcoma, undifferentiated high-grade pleomorphic sarcoma, pleomorphicsarcoma with prominent inflammation, pleomorphic sarcoma with giant cells, malignant fibrous histiocytoma (including storiform-pleomorphic and inflammatory subtypes), fibrosarcoma, and myxofibrosarcoma (located deep to the fascia in muscle). Radiation therapy with three cycles of pembrolizumab will be administered as neoadjuvant therapy for patients randomized to the experimental arm. These patients will also receive up to fourteen cycles of adjuvant pembrolizumab after surgical resection. Patients in the standard of care arm will receive neoadjuvant radiotherapy (50 Gy in 25 fractions) followed by surgical resection as in RTOG 0630.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 12 years
* Histologically confirmed diagnosis of grade 2 or 3 out of 3 UPS or dedifferentiated/pleomorphic LPS of the extremity (including limb girdle, i.e. shoulder or hip) that measures greater than 5 cm in any direction as assessed by imaging
* Patients with non-melanomatous skin cancer, in situ carcinoma, or low-risk prostate cancer can be enrolled.
* ECOG Performance Status of 0 or 1
* Resectable primary tumor with no evidence of metastatic disease by imaging.
* Adequate organ function within 10 days of Day 1
* Written, voluntary informed consent
* Fertile men and women of childbearing potential must agree to use an effective method of birth control from Day 1 of study and for 120 days after last pembrolizumab administration in both sexes. Women of childbearing potential include pre-menopausal women and women within the first 2 years of the onset of menopause. Women of childbearing potential must have a negative pregnancy test ≤ 72 hours prior to Day 1 of study.

Exclusion Criteria:

* Prior chemotherapy, targeted small molecule therapy, or radiation therapy for current diagnosis of sarcoma
* Prior radiation therapy in excess of 20 Gy to the site of the current diagnosis of sarcoma. No overlap with prior radiation fields in excess of 20 Gy is allowed.
* Concurrent, clinically significant, active malignancies within two years of study enrollment.
* Patients with locally recurrent sarcoma after surgery alone are eligible for enrollment if other inclusion criteria are met.
* Patients with severe and/or uncontrolled concurrent medical disease that in the opinion of the investigator could cause unacceptable safety risks or compromise compliance with the protocol
* Major surgery within four weeks prior to Day 1 of study or who have not recovered adequately from prior surgery.
* Currently receiving a study therapy or if they had an investigational agent within 4 weeks at the time of enrollment.
* Women who are pregnant or nursing/breastfeeding, or expecting to conceive or men who are expecting to father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of pembrolizumab.
* Inability to comply with protocol required procedures
* Diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy by oral or IV routes within 7 days prior to the first dose of trial treatment
* Known history of active TB (Bacillus Tuberculosis)
* Hypersensitivity to pembrolizumab or any of its excipients
* Metastatic disease or regional lymph node involvement. Chest CT will be mandatory prior to enrollment to evaluate for the presence of metastatic disease. Pulmonary nodule(s) < 5 mm without a histological diagnosis may not be the basis for study exclusion given the lack of specificity of chest CT. If pulmonary nodule(s) measuring 6 - 10 mm are noted on chest CT but appear stable relative to prior chest imaging of at least 6 months duration or if 18FDG-PET scan indicates that the nodule(s) are unlikely to be metastatic disease, then this is permitted. Pulmonary nodules >10 mm should be considered metastatic unless proven otherwise by biopsy/resection or stable appearance for at least 6 months on imaging.
* Unresectable disease or medically inoperable
* Planned to receive neoadjuvant or adjuvant chemotherapy for current diagnosis of localized soft tissue sarcoma
* Active autoimmune disease that has required systemic treatment in the past two years (i.e. with use of disease modifying agents, systemic corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Has a history of (non-infectious) pneumonitis that required systemic steroids or current pneumonitis.
* Active infection requiring systemic therapy
* Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent
* Known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies)
* Known active Hepatitis B (e.g., HBsAg reactive, confirmed by detectable viral load) or Hepatitis C (e.g., HCV RNA [qualitative] detected)
* Received a live vaccine within 30 days of planned start of study therapy. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.
* Diagnosis of scleroderma.
* Diagnosis of inflammatory bowel disease (Crohn's disease or Ulcerative Colitis).

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2017-07-19 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Disease free survival | 2 Years
  Disease recurrence is defined as clinically diagnosed or biopsy-confirmed recurrent sarcoma at a site distant to the primary tumor, including nodal metastasis, loco-regional recurrence, and death without documented recurrence.

SECONDARY OUTCOMES:
Loco-regional disease-free survival | 5 years
  The length of time after treatment ends without any locoregional recurrence of sarcoma.
Distant disease free survival | 5 years
  The length of time after treatment ends that the patient survives without any signs or symptoms of sarcoma
Overall survival | 5 years
  The length of time from the start of treatment that patients diagnosed with sarcoma are still alive.
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 5 years
  Test the safety of neoadjuvant pembrolizumab administered with conventionally fractionated radiotherapy targeting soft tissue sarcoma of the extremity.

CONTACTS AND LOCATIONS:
Overall Officials: David Kirsch, MD, PhD, Principal Investigator — Princess Margaret Cancer Center
Locations (20):
- United States (15):
  - University of California Los Angeles, Los Angeles, California
  - Mayo Clinic- Florida, Jacksonville, Florida
  - University of Iowa Hospitals & Clinics, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Johns Hopkins University, Baltimore, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Washington University, St Louis, Missouri
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke University, Durham, North Carolina
  - The Ohio State University, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - University of Pennsylvania- Abramson Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh (UPMC Hillman Cancer Center), Pittsburgh, Pennsylvania
- Australia (3):
  - Chris O'Brien Hospital, Camperdown, New South Wales
  - Princess Alexandra Hospital, Brisbane, Queensland
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
- McGill University Health Centre, Montreal, Quebec, Canada
- Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mowery YM, Ballman KV, Hong AM, Schuetze SM, Wagner AJ, Monga V, Heise RS, Attia S, Choy E, Burgess MA, Bae S, Pryor DI, Van Tine BA, Tinoco G, Chmielowski B, Freeman C, Gronchi A, Meyer CF, Dickson MA, Hartner L, Davis LE, Powers BC, Moding EJ, Weinhold KJ, van de Rijn M, Brigman BE, Riedel RF, Kirsch DG. Safety and efficacy of pembrolizumab, radiation therapy, and surgery versus radiation therapy and surgery for stage III soft tissue sarcoma of the extremity (SU2C-SARC032): an open-label, randomised clinical trial. Lancet. 2024 Nov 23;404(10467):2053-2064. doi: 10.1016/S0140-6736(24)01812-9. Epub 2024 Nov 12. PMID 39547252